CLINICAL TRIAL: NCT05511324
Title: Simulation-Based Caregiving Skills Training for Family Members of High Grade Glioma Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-0377; NCI-2022-07002 (Other: NCI-CTRP Clinical Trials Reporting Registry); R21CA273782 (NIH)
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline Assessment (Other): Participants will be asked to complete a baseline assessment of questionnaires that will ask:
  * Demographic information (such as your age, sex, and race)
  * Psychological and physical health
  Interventions: Behavioral: Questionnaires
- Caregiver Intervention Sessions (Other): Caregiver will take part in 4 caregiver intervention sessions. The first 2 sessions will take place in the Simulation Center at the hospital when you are scheduled for treatment or a follow-up appointment. The remaining 2 sessions will be done remotely using a videoconference platform (such as Zoom) and will focus on discussing your caregiver's role and experiences and suggesting coping and self-care strategies.
  Interventions: Behavioral: Caregiver Assessment

INTERVENTIONS:
Behavioral: Questionnaires — Participants will be asked to complete this assessment on your own time, and it should take about 40 minutes.
  Arms: Baseline Assessment
Behavioral: Caregiver Assessment — These sessions will involve simulation-based, caregiving skill training, and your caregiver will be taught skills to help support you (such as feeding, hygiene, mobility, medication administration, and care coordination).
  Arms: Caregiver Intervention Sessions

SUMMARY:
Family caregivers of patients with a primary brain tumor experience a high caregiving load including assistance with activities of daily living without any formal training. It is not surprising that this vulnerable caregiver population reports high levels of distress along with numerous caregiving-related concerns, which may compromise their ability to provide quality care. This project will examine the feasibility and initial evidence for efficacy of a caregiving skills intervention aiming to improve caregiver and patient psychological health; caregiving efficacy and role adjustment; and reduce patient cancer-related symptoms and healthcare utilization.

DETAILED DESCRIPTION:
Trial 1 (single-arm study)

• Aim 1: Examine the usability of the intervention content and trial assessments in 10 caregiver-patient dyads to refine study procedures as needed.

Trial 2 (RCT)

Aim 1 (primary aim): Determine the feasibility of implementing a caregiving intervention using a randomized controlled design in 50 caregiver-HGG patient dyads.

Aim 2: Evaluate the initial evidence for intervention efficacy relative to a WLC group regarding patient and caregiver psychological symptoms (primary outcome), caregiver caregiving efficacy and role adjustment, and patient cancer-related symptoms and healthcare utilization (secondary outcomes).

Aim 3: Understand caregivers' experiences using qualitative methods regarding participation in this study and explore emerging themes as possible intervention mediators/moderators to be examined in future research.

ELIGIBILITY:
Inclusion Criteria:

* FCGs (e.g., spouse/partner, parent, adult child) of patients diagnosed with HGG receiving any form of cancer treatment (including palliative intent) at MDACC.
* Patients must have a Karnofsky Performance Status (KPS) of 100 to 50. If the patient's Karnofsky Performance Status drops below 50 both patient and caregiver will be removed from the study.
* Both FCGs and patients must be willing to participate and (1) ≥18 years old and able to (2) read and speak English and (3) provide informed consent.

Exclusion Criteria:

* FCGs who regularly participate in psychotherapy with a licensed professional (self-reported).
* Patients with cognitive impairment that would impede ability to complete self-report surveys as documented in the medical record.
* Children under the age of 18 will not be included in this trial. First and foremost, it is unlikely that a person under the age 18 is diagnosed with an HGG.
* Childhood brain tumors tend to be diagnosed in infancy and the caregiving and symptom management needs are vastly different than in the adult patient population. Additionally, the assessment tools are not validated for minors.
* While pregnant caregivers (self-reported) are study eligible, we will also exclude pregnant patients (medical notes). It is unlikely that patients diagnosed with an HGG will be pregnant. Moreover, the current caregiver intervention is not designed to address the care needs of pregnant cancer patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
M. D. Anderson Symptom Inventory (MDASI) questionnaires | through study completion and average of 1 year.
  M. D. Anderson Symptom Inventory (MDASI) questionnaires score scale ranges ( 0-10) 0 has not been present been and 10 is bad as you can imagine.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Milbury, MA,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2025-01-29): https://cdn.clinicaltrials.gov/large-docs/24/NCT05511324/ICF_000.pdf